CLINICAL TRIAL: NCT01018706
Title: Goodness of Clinical History During Stemi PCI (GHOST)
Brief Title: Goodness of Clinical History During Stemi PCI
Acronym: GHOST
Status: Completed | Type: Observational
Sponsor: Umberto I Hospital, Frosinone Italy (Other)
Responsible Party: Principal Investigator, Menichelli Maurizio, Director of Cardiology Division, Umberto I Hospital, Frosinone Italy
Other Study IDs: GHOST
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Myocardial Infarction
Keywords: Primary pci; Stent; Medical Hystory; Antiplatelet therapy; Compliance
MeSH Terms: conditions — Myocardial Infarction; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI patients treated with PCI: Four hundred patients with STEMI treated with primary PCI or rescue PCI.

SUMMARY:
The purpose of this study is to confirm or confute the hypothesis that in patients treated with primary pci is not always possible to collect an adequate medical history, the investigators created a clinical registry in which the investigators collect current or previous medical history relevant to DES utilization , in two distinct times.

DETAILED DESCRIPTION:
GHOST Registry

Use of drug-eluting stent (DES) in STEMI is sometimes limited, by the concern that adequate information, relating to the current or previous medical history, can not be obtained due to the patient's critical condition. A less than adequate medical history would expose patients treated with DES to a particular risk in case that an absolute or relative contraindication to the required long-term double antiplatelet therapy is not fully elucidated before DES implantation.

To confirm or confute the hypothesis that in patients treated with primary pci is not always possible to collect an adequate medical history, we created a clinical registry in which we collect current or previous medical history relevant to DES utilization , in two distinct times:

Time zero in which the medical history collection is taken in the cath-lab during the primary pci

Time one in which the second medical history collection is taken 4 days after the index procedure when the patient clinical conditions no longer impede an adequate medical history collection.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients presenting with STEMI treated with primary or rescue PCI

Exclusion Criteria:

* Patient in cardiogenic shock and all those patients unable to communicate with the doctors at the moment of medical history taking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four hundred patients with STEMI treated with primary PCI or rescue PCI.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Adequacy of medical history collection at the moment of primary pci and 4 days after the index procedure | Adequacy of medical history collection at the moment of primary pci and 4 days after the index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Interventional cardiology divisione , Umberto I Hospital, Frosinone, Frosinone, Italy